CLINICAL TRIAL: NCT05566652
Title: Neural Pressure Support for Low Pulmonary Compliance
Acronym: NPS_LowCrs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Full Professor, Policlinico Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NPS
Record Dates: First submitted 2022-09-13; First posted 2022-10-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Acute Respiratory Failure
Keywords: NPS; WOB; AI

STUDY DESIGN:
Intervention Model Description: This is an interventional prospective crossover physiological study that will take place at the Intensive Care Unit "E. Vecla", Department of Anesthesia, Intensive Care and Emergency, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPS (Experimental): To evaluate WOB and asynchronies in patients with low respiratory system compliance undergoing Neural Pressure Support Ventilation.
  Interventions: Device: Neural Pressure Support; Drug: Pressure Support Ventilation
- PSV (Sham Comparator): To evaluate WOB and asynchronies in patients with low respiratory system compliance undergoing Pressure Support Ventilation.
  Interventions: Device: Neural Pressure Support; Drug: Pressure Support Ventilation

INTERVENTIONS:
Device: Neural Pressure Support — To evaluate WOB and asynchronies in patients with low respiratory system compliance undergoing either PSV and NPS.
Drug: Pressure Support Ventilation — To evaluate WOB and asynchronies in patients with low respiratory system compliance undergoing either PSV and NPS.

SUMMARY:
With this interventional prospective study, we aim at comparing the effectiveness of Neural Pressure Support (NPS) in reducing respiratory work and patient-ventilator asynchronies as compared with standard Pressure Support Ventilation (PSV), in a cohort of patients with Acute Respiratory Failure (ARF) and low respiratory system compliance.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is a critical condition caused by impaired function of the lungs.1,2 The cornerstone of ARF management is invasive mechanical ventilation (IMV).3,4 Unfortunately, despite lifesaving, IMV is associated with several side effects (e.g., ventilator-associated pneumonia, ventilator associate induced lung injury, diaphragmatic dysfunction), and thus liberation from invasive mechanical ventilation is an everyday effort for critical care physicians.5

Pressure support ventilation (PSV) is one of the most widely used mechanical ventilation modes for liberation from IMV.6 PSV is a partial ventilatory mode: the ventilator and the patient co-operate to generate the inspiratory and expiratory pressures, flows, and volumes. During conventional PSV, the initiation of the breath is triggered by a reduction in expiratory pressure or a drop in expiratory flow.7 The termination of the breath occurs when the inspiratory flow falls to a predetermined fraction of the peak inspiratory flow.8

The main goal of mechanical ventilation is to help restore gas exchange and reduce the work of breathing (WOB) by assisting respiratory muscle activity.9 Knowing the determinants of WOB is essential for the effective use of mechanical ventilation and also to assess patient readiness for weaning. To reduce WOB, PSV needs to be synchronous and smooth interaction should happen between the ventilator and the respiratory muscles.10

Ideally, the ventilator trigger and cycling should coincide with the beginning and end of the patient's inspiratory effort.11 However, patient-ventilator asynchrony is common during PSV,12,13 thereby contributing to an increased work of breathing and an increased duration of mechanical ventilation.14

An important objective of assisted or patient-triggered mechanical ventilation is to avoid ventilator-induced diaphragmatic dysfunction by allowing the patient to generate spontaneous efforts.15 A second objective is to reduce the patient's work of breathing by delivering a sufficient level of ventilatory support.16 Finally, intuition suggests that a good match between patient respiratory efforts and ventilator breaths optimizes patient comfort and reduces work of breathing.17 Patient-ventilator asynchrony can be defined as a mismatch between the patient and ventilator inspiratory and expiratory times.18 Although inspiratory and expiratory delays are almost inevitable with most ventilatory modes, several patterns of major asynchrony exist and can be easily detected by clinicians.14

The diaphragmatic electrical activity (EAdi) can be used to optimize the ventilator settings and improve the matching between patient and ventilator. The EAdi signal is a surrogate of respiratory brain stem output and can be recorded using specialized nasogastric tubes equipped with electrodes.19

The Neural Pressure Support (NPS) is a newer ventilation mode that includes neural trigger and termination of inspiration based on the electrical activity of the diaphragm (Edi). NPS delivers a constant airway pressure support independent of the patient's efforts.20

The NPS may be particularly beneficial for ARF patients with lower respiratory compliance. Indeed, in this cohort, during standard PSV, expiratory cycling may be hampered by several asynchronies.21 However, to our knowledge, the effectiveness of NPS in reducing asynchronies and respiratory work has not been tested and compared with standard PSV in patients with low respiratory system compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admission to Intensive Care Unit (ICU) for ARF
* Low compliance of the respiratory system (Crs ≤ 30 ml/cmH2O)
* Written informed consent obtained

Exclusion Criteria:

* Contraindication to nasogastric tube insertion (gastroesophageal surgery in the previous 3 months, gastroesophageal bleeding in the previous 30 days, history of esophageal varices, facial trauma)
* Increased risk of bleeding with nasogastric tube insertion, due to severe coagulation disorders and severe thrombocytopenia ( i.e., International Normalized Ratio (INR) > 2 and platelets count < 70.000/mm3)
* Severe hemodynamic instability (noradrenaline > 0.3 μg/kg/min and/or use of vasopressin)
* Failure to obtain a stable EAdi signal
* Central nervous system or neuromuscular disorders
* Moribund status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Work Of Breathing (WOB) | 30 minutes ventilatory traces recording
  We hypothesize that Neural Pressure Support (NPS) is able to improve the patient-ventilator interaction, thus reducing significantly the patient's work of breathing (WOB). WOB will be evaluated by the off-line analysis of the esophageal pressure waveform.

SECONDARY OUTCOMES:
Asynchronies | 30 minutes ventilatory traces recording
  We hypothesize that Neural Pressure Support (NPS) is able to improve the patient-ventilator interaction, thus reducing significantly the asynchronies between patient and ventilator. Asynchronies will be estimated by the Asynchrony Index (AI) calculated off-line by ventilatory waveforms analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
According to the International Council for Harmonisation of Technical Requirements (ICH) guidelines for the Good Clinical Practice (GCP), the monitoring team must check the Case Report Form (CRF) entries against source documents. The personnel bound by professional secret, must maintain the confidentiality of all personal identity or personal medical information. The confidentiality of records that could identify subjects should be protected, only initials of the name and the first name will be registered with a inclusion coded number for the study (no name nor address nor identifying data).
  Paper-based CRF will be designed by the PI. A unique code will be assigned to each participant in order to de-identify the data. It is the Investigator's responsibility to ensure the accuracy of all data entered and recorded in the CRFs.
  The database will be password protected and stored on a password-protected Personal Computer in a research office in the critical care department.

REFERENCES:
- [Background] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Background] Meyer NJ, Gattinoni L, Calfee CS. Acute respiratory distress syndrome. Lancet. 2021 Aug 14;398(10300):622-637. doi: 10.1016/S0140-6736(21)00439-6. Epub 2021 Jul 1. PMID 34217425
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Pelosi P, Ball L, Barbas CSV, Bellomo R, Burns KEA, Einav S, Gattinoni L, Laffey JG, Marini JJ, Myatra SN, Schultz MJ, Teboul JL, Rocco PRM. Personalized mechanical ventilation in acute respiratory distress syndrome. Crit Care. 2021 Jul 16;25(1):250. doi: 10.1186/s13054-021-03686-3. PMID 34271958
- [Background] Fan E, Del Sorbo L, Goligher EC, Hodgson CL, Munshi L, Walkey AJ, Adhikari NKJ, Amato MBP, Branson R, Brower RG, Ferguson ND, Gajic O, Gattinoni L, Hess D, Mancebo J, Meade MO, McAuley DF, Pesenti A, Ranieri VM, Rubenfeld GD, Rubin E, Seckel M, Slutsky AS, Talmor D, Thompson BT, Wunsch H, Uleryk E, Brozek J, Brochard LJ; American Thoracic Society, European Society of Intensive Care Medicine, and Society of Critical Care Medicine. An Official American Thoracic Society/European Society of Intensive Care Medicine/Society of Critical Care Medicine Clinical Practice Guideline: Mechanical Ventilation in Adult Patients with Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 May 1;195(9):1253-1263. doi: 10.1164/rccm.201703-0548ST. PMID 28459336
- [Background] Hess DR. Ventilator waveforms and the physiology of pressure support ventilation. Respir Care. 2005 Feb;50(2):166-86; discussion 183-6. PMID 15691390
- [Background] Spahija J, de Marchie M, Albert M, Bellemare P, Delisle S, Beck J, Sinderby C. Patient-ventilator interaction during pressure support ventilation and neurally adjusted ventilatory assist. Crit Care Med. 2010 Feb;38(2):518-26. doi: 10.1097/CCM.0b013e3181cb0d7b. PMID 20083921
- [Background] MacIntyre NR. Clinically available new strategies for mechanical ventilatory support. Chest. 1993 Aug;104(2):560-5. doi: 10.1378/chest.104.2.560. No abstract available. PMID 8339649
- [Background] Nava S, Bruschi C, Rubini F, Palo A, Iotti G, Braschi A. Respiratory response and inspiratory effort during pressure support ventilation in COPD patients. Intensive Care Med. 1995 Nov;21(11):871-9. doi: 10.1007/BF01712327. PMID 8636518
- [Background] Leung P, Jubran A, Tobin MJ. Comparison of assisted ventilator modes on triggering, patient effort, and dyspnea. Am J Respir Crit Care Med. 1997 Jun;155(6):1940-8. doi: 10.1164/ajrccm.155.6.9196100.
- [Background] Yamada Y, Du HL. Analysis of the mechanisms of expiratory asynchrony in pressure support ventilation: a mathematical approach. J Appl Physiol (1985). 2000 Jun;88(6):2143-50. doi: 10.1152/jappl.2000.88.6.2143. PMID 10846029
- [Background] Tokioka H, Tanaka T, Ishizu T, Fukushima T, Iwaki T, Nakamura Y, Kosogabe Y. The effect of breath termination criterion on breathing patterns and the work of breathing during pressure support ventilation. Anesth Analg. 2001 Jan;92(1):161-5. doi: 10.1097/00000539-200101000-00031. PMID 11133620
- [Background] Tassaux D, Gainnier M, Battisti A, Jolliet P. Impact of expiratory trigger setting on delayed cycling and inspiratory muscle workload. Am J Respir Crit Care Med. 2005 Nov 15;172(10):1283-9. doi: 10.1164/rccm.200407-880OC. Epub 2005 Aug 18. PMID 16109983
- [Background] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Background] Vassilakopoulos T, Petrof BJ. Ventilator-induced diaphragmatic dysfunction. Am J Respir Crit Care Med. 2004 Feb 1;169(3):336-41. doi: 10.1164/rccm.200304-489CP. No abstract available. PMID 14739134
- [Background] Brochard L, Harf A, Lorino H, Lemaire F. Inspiratory pressure support prevents diaphragmatic fatigue during weaning from mechanical ventilation. Am Rev Respir Dis. 1989 Feb;139(2):513-21. doi: 10.1164/ajrccm/139.2.513. PMID 2643905
- [Background] Sassoon CS, Foster GT. Patient-ventilator asynchrony. Curr Opin Crit Care. 2001 Feb;7(1):28-33. doi: 10.1097/00075198-200102000-00005. PMID 11373508
- [Background] Tobin MJ, Jubran A, Laghi F. Patient-ventilator interaction. Am J Respir Crit Care Med. 2001 Apr;163(5):1059-63. doi: 10.1164/ajrccm.163.5.2005125. No abstract available. PMID 11316635
- [Background] Dres M, Demoule A. Monitoring diaphragm function in the ICU. Curr Opin Crit Care. 2020 Feb;26(1):18-25. doi: 10.1097/MCC.0000000000000682. PMID 31876624
- [Background] Liu L, Xu XT, Yu Y, Sun Q, Yang Y, Qiu HB. Neural control of pressure support ventilation improved patient-ventilator synchrony in patients with different respiratory system mechanical properties: a prospective, crossover trial. Chin Med J (Engl). 2021 Jan 19;134(3):281-291. doi: 10.1097/CM9.0000000000001357. PMID 33470654
- [Background] Mirabella L, Cinnella G, Costa R, Cortegiani A, Tullo L, Rauseo M, Conti G, Gregoretti C. Patient-Ventilator Asynchronies: Clinical Implications and Practical Solutions. Respir Care. 2020 Nov;65(11):1751-1766. doi: 10.4187/respcare.07284. Epub 2020 Jul 14. PMID 32665426